CLINICAL TRIAL: NCT02004158
Title: Study of a Positive Psychology Program to Improve Healthy Behaviors After an Acute Coronary Syndrome: Proof of Concept Study
Brief Title: Positive Psychology to Improve Healthy Behaviors After an Acute Coronary Syndrome
Acronym: PEACE II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Jeff C. Huffman, MD, Director, Cardiac Psychiatry Research Program, Massachusetts General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2013P001961; 1R01HL113272-01A1 (NIH)
Record Dates: First submitted 2013-12-03; First posted 2013-12-06 (Estimated); Results first posted 2017-07-24 (Actual); Last update posted 2017-07-24 (Actual); Status verified 2017-05

CONDITIONS: Acute Coronary Syndrome
Keywords: Acute coronary syndrome; Health behavior; Mental health
MeSH Terms: conditions — Acute Coronary Syndrome; Health Behavior; Psychological Well-Being

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Positive psychology (Experimental): Positive psychology intervention
  Interventions: Behavioral: Positive psychology intervention

INTERVENTIONS:
Behavioral: Positive psychology intervention

SUMMARY:
In this proof-of-concept study, the investigators will assess the ease and usefulness of a positive psychology program in patients with acute coronary syndrome and less-than-optimal adherence to health behaviors. The investigators believe that positive psychology (a field that studies boosting positive emotions rather than simply reducing negative emotions) will help this cardiac population to be more healthy. The investigators want to determine whether this positive psychology program has the potential to be an adjunctive treatment for cardiac populations.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients admitted to one of three cardiac inpatient units at Massachusetts General Hospital.
* Primary diagnosis of acute coronary syndrome (myocardial infarction or unstable angina).
* Less-than-optimal adherence to health behaviors. This will be defined as a mean score of less than 15 on the Medical Outcomes Study Specific Adherence Scale (scores range from 3-18, with higher scores indicating better adherence).

Exclusion Criteria:

* Cognitive deficits, assessed via a 6-item cognitive screen used to assess appropriate participation of medically-ill patients in research studies.
* Patients not prescribed aspirin at discharge.
* Inability to communicate in English.
* Inability to participate in physical activity.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Huffman, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Positive Psychology
Started | 23
Completed | 20
Not Completed | 3

BASELINE CHARACTERISTICS:
Arm/Group | Positive Psychology
Number analyzed (Participants) | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.4 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 12
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 18
  More than one race | 1
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Rate of Exercise Completion
Description: Rate of exercise completion will be measured by the number of participants who have a good rate of completion of exercises. There are 8 exercises in total. A good rate of completion will be defined as an average of 5 or more exercises completed per subject.
Time Frame: 8 weeks
Measure: Number; unit: Participants
Arm/Group | Positive Psychology
Number analyzed (Participants) | 23
Participants | 17

2. Primary Outcome: Ease of Exercises
Description: Ease of exercises will be measured by a self-report 10-point Likert scale (0=not easy to complete, 10=very easy to complete). Ease will be defined as an average score of 6 or more on this scale.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Positive Psychology
Number analyzed (Participants) | 23
scores on a scale | 7.4 (2.1)

3. Primary Outcome: Self-reported Psychological Impact of Exercises
Description: Psychological impact of exercises will be measured by two self-reported 10-point Likert scales. One scale measures optimism after completing the exercise (0=not optimistic, 10=very optimistic), and the other scale measures happiness after completing the exercise (0=not happy, 10=very happy). Psychological impact will be defined as an average score of 6 or more on both of these scales.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: points
Arm/Group | Positive Psychology
Number analyzed (Participants) | 23
points
  Optimism | 7.9 (1.5)
  Happiness | 8.0 (1.6)

4. Secondary Outcome: Objective Psychological Impact of Exercises
Description: Object psychological impact of exercises will be measured by clinician-administered questionnaires given at baseline and again at 8 weeks. These questionnaires include:
  1. Life Orientation Test-Revised (scores range from 6-30; a high score means higher optimism)
  2. Positive and Negative Affect Schedule (scores range from 10-50; a higher score means higher levels of affect)
  3. Hospital Anxiety and Depression Scale (scores range from 0-42; a high score means higher depression and anxiety).
  Objective psychological impact will be defined as having significantly improved scores at 8 weeks as compared to scores at baseline.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: points
Groups:
- Positive Psychology: Positive psychology intervention (Baseline data)
- Positive Psychology: Positive psychology intervention (8 week data)
Arm/Group | Positive Psychology | Positive Psychology
Number analyzed (Participants) | 20 | 20
points
  LOT-R | 23.5 (4.8) | 23.0 (5.8)
  PANAS | 35.1 (7.9) | 38.2 (8.6)
  HADS | 13.4 (8.9) | 9.0 (5.6)

ADVERSE EVENTS:
Time Frame: 11 months (duration of study)
Arm/Group | Positive Psychology
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes